CLINICAL TRIAL: NCT00309582
Title: Plasma Nevirapine Levels and Adverse Events Among HIV-Infected Patients Concurrently Receiving Nevirapine-Based Antiretroviral Therapy and Fluconazole
Brief Title: Nevirapine Levels and Fluconazole
Status: Completed | Type: Observational
Sponsor: Bamrasnaradura Infectious Diseases Institute (Other Government)
Other Study IDs: BIR2405
Record Dates: First submitted 2006-03-30; First posted 2006-04-03 (Estimated); Last update posted 2006-04-03 (Estimated); Status verified 2005-11

CONDITIONS: Nevirapine; Fluconazole; Adverse Event

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Nevirapine (NVP)-based antiretroviral therapy (ART) has been commonly used in many developing countries due to its affordability and feasibility. Nonetheless, the potential drug-drug interaction between NVP and fluconazole (FLU) is a major concern. NVP can induce cytochrome P450 isoenzymes in the liver while FLU inhibit the activity of this enzyme. The recent report has demonstrated that fluconazole significantly raises plasma NVP levels and may cause serious hepatotoxicity. Conversely, NVP does not significantly influence the plasma level of FLU. However, there have not been enough data or any recommendations to adjust NVP dosage for the concurrent use of both drugs in order to avoid the adverse events. A previous study has demonstrated that genetic disposition may play a role in NVP hypersensitivity reactions. There is little data of safety and tolerability for concurrent use of NVP and FLU in Asian populations. We therefore conducted this prospective observational study to compare the trough plasma NVP levels and frequencies of adverse events among antiretroviral HIV-infected patients who did not receive FLU and received FLU in different dosages for cryptococcosis prophylaxis or treatment; and subsequently received NVP-based ART regimens.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected patients >15 years of age,
2. naïve to antiretroviral therapy,
3. were initiated with a NVP-based ART regimen,
4. used NVP 200-mg once-daily lead-in dose, prior to escalation to 200 mg twice daily.

Exclusion Criteria:

1. creatinine level was higher than 2.0 mg/ml
2. liver aminotransferase enzyme was higher than five times of upper normal limit
3. receiving a medication that has drug-drug interactions with NVP or FLU

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Weerawat Manosuthi, MD, Principal Investigator — Bamrasnaradura Infectious Diseases Institute